CLINICAL TRIAL: NCT06013930
Title: Exploring the Efficacy of Alternative Treatments for Depression and Anxiety Among College Students: A Randomized Control Trial
Brief Title: Exploring the Efficacy of Treatments for Anxiety and Depression Among College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Dakota (Other)
Collaborators: Subtle Energy Funders Collective (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-247
Record Dates: First submitted 2023-04-19; First posted 2023-08-28 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either: 1) External Qigong, 2) Mindfulness Meditation, or 3) Psychoeducation.
Who Masked: Outcomes Assessor
Masking Description: The PI will randomly assign participants to condition and coordinate treatment group scheduling; the assessor will be blinded to condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- External Qigong (Experimental): Participants will meet individually with the Qigong practitioner once a week for three weeks for 30-minute segments.
  Interventions: Behavioral: External Qigong
- Mindfulness Meditation (Experimental): Participants will meet individually with the mindfulness practitioner once a week for three weeks for 30-minute segments.
  Interventions: Behavioral: Mindfulness Meditation
- Psychoeducation (Active Comparator): In the psychoeducation arm, participants will receive recordings online, once a week for three weeks which will be approximately 30 minutes in length.
  Interventions: Other: Psychoeducation

INTERVENTIONS:
Behavioral: External Qigong — External Qigong will be facilitated by a seasoned Qigong practitioner. The Qigong practitioner will assist participants in learning how to use the healing powers of their bodies to decrease feelings of anxiety and/or depression
  Arms: External Qigong
Behavioral: Mindfulness Meditation — Mindfulness meditation will be facilitated by a seasoned mindfulness practitioner. Participants will be guided through a meditation designed to help increase a sense of interconnectedness among their college community. They will also learn how to deconstruct feelings of anxiety and/or depression into sensory, emotional, cognitive, and behavioral components.
  Arms: Mindfulness Meditation
Other: Psychoeducation — In the psychoeducation arm, participants will receive information related to managing anxiety and/or depression through a recorded presentation. Participants will learn about stress-management techniques to help reduce symptoms of anxiety and/or depression. They will also receive information on resources that could be helpful in treating anxiety and/or depression.
  Arms: Psychoeducation

SUMMARY:
The goal of this randomized control group is to learn about effective treatments for college students experiencing anxiety and/or depression. The main questions this clinical trial aims to answer are: 1) Can alternative treatments decrease anxiety and/or depression among college students? 2) Can alternative treatments increase retention rates among college students experiencing anxiety and/or depression?

Participants will be randomly assigned to one of three intervention groups: external qigong, mindfulness meditation, or psychoeducation. Researchers will compare outcomes from each group to explore treatment differences.

DETAILED DESCRIPTION:
Method/Design. This study will be a single-site, three-arm, randomized, controlled trial. College students (N=51) with elevated depression and/or anxiety will be randomized to either external qigong (EQ), mindfulness meditation (MM), or psychoeducation (PE). Each intervention will be applied for 30 minutes, once a week for three weeks in a community setting. The co-primary outcomes, depression and anxiety, and the secondary outcome, intention to persist in college, will be assessed by a blinded researcher at baseline, one-week post treatment, and one-month follow-up. Change in sense of connection during the treatment session, measured with a comprehensive battery of self-report indices, will be the primary therapeutic mechanism.

Aims and Objectives. The proposed project's central hypothesis is that EQ will increase students' mental health and intention to persist in college by balancing the flow of energy in their bodies. Aim 1. Examine EQ's acceptability in a sample of college students with depression and/or anxiety. Hypothesis: Student retention (i.e., attendance in both treatment sessions) and self-reported treatment acceptability will be better for EQ relative to PE. EQ and MM will demonstrate equivalent acceptability. Aim 2. Determine EQ's effect on anxiety, depression (co-primary outcomes), and intention to persist in college (secondary outcome) over time. Hypothesis: EQ will decrease depression and anxiety while increasing intention to persist in college relative to PE from baseline to one-month follow-up. The co-primary and secondary outcome scores will not differ between EQ and MM. Aim 3. Investigate EQ's immediate effect on students' sense of connection (therapeutic mechanism). Hypothesis: EQ will increase students' sense of connection relative to PE during the treatment sessions. EQ and MM will have equivalent effects on sense of connection.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Currently enrolled in a two or four-year college.
* English speaking.
* Willing to travel to the study location.
* Access to a computer or smartphone with a Wifi connection.
* Score of a three or higher on the Generalized Anxiety Disorder 2-item and/or score of a three or higher on the Patient Health Questionnaire-2.

Exclusion Criteria:

* Not currently enrolled in college.
* Not able to travel to the study location.
* No access to a computer or smartphone with Wifi.
* Score < 3 on the Generalized Anxiety Disorder-2 and < 3 on the Patient Health Questionnaire-2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Anxiety | Change from baseline assessment, post treatment (one week after the final treatment session), and follow-up (one month after the final treatment session).
  Symptoms of anxiety will be assessed through a trait anxiety assessment (State-Trait-Anxiety Inventory). The range of possible scores spans from a minimum score of 20 to a maximum score of 80 - the higher the score, the higher the symptoms of anxiety.
Depression | Change from baseline assessment, post treatment (one week after the final treatment session), and follow-up (one month after the final treatment session).
  Symptoms of depression will be assessed through a trait depression assessment (Beck Depression Inventory). Scores from the Beck Depression Inventory range from 0-63, with higher scores representing high depression levels.

SECONDARY OUTCOMES:
Intention to persist in college | Baseline, post treatment (one week after the final treatment session), and follow-up (one month after the final treatment session).
  Change in participants' intention to persist in college will be assessed through an individual item rated in a numeric rating scale. Scores range from 0 to 5 with higher scores reflecting greater intent to remain in college.
Anxiety | Changes in participant's state anxiety will be captured within 5-minutes prior to each intervention and within 5 minutes after each intervention (mindfulness, external qigong, and psychoeducation).
  Symptoms will be assessed through a state anxiety assessment. Scores range from 0-60 with higher scores indicating higher levels of anxiety.
Depression | Changes in participant's state depression will be captured within 5-minutes prior to each intervention and within 5 minutes after each intervention (mindfulness, external qigong, and psychoeducation).
  Symptoms will be assessed through a state depression assessment. Scores range from 0-20 with higher scores indicating higher levels of depression.

OTHER OUTCOMES:
Adverse Childhood Experiences questionnaire. | Baseline
  Participants adverse childhood experiences will be assessed at baseline to explore how childhood adversities moderate outcomes.The ACEs questionnaire was adapted from the Felitti et al., (1998) wave two survey and current questions used by the CDC's telephone Behavioral Risk Factor Surveillance System survey collected in all 50 states. ACES range between 0-13 and the higher the score, the higher the number of ACES.
Sensation Manikin | Changes in participant's state body sensations will be captured within 5-minutes prior to each intervention and within 5 minutes after each intervention (mindfulness, external qigong, and psychoeducation).
  Change in the distribution of pleasant and unpleasant bodily sensations. Scores can range from 0-100 for pleasant (higher scores indicate higher pleasant feelings) and 0-100 for unpleasant feelings (higher scores indicate higher levels of unpleasant sensations).
Trait Self-Transcendence | Baseline, post treatment (one week after the final treatment session), and follow-up (one month after the final treatment session).
  Change in trait self-transcendence from baseline through 3-month follow-up will be assessed with the Nondual Awareness Dimensional Assessment - Trait Version. Scores range from 0 to 52, with higher scores reflecting greater trait self-transcendence.
Self-Transcendent State | Changes in participant's self-transcendence will be captured within 5-minutes prior to each intervention and within 5 minutes after each intervention (mindfulness, external qigong, and psychoeducation).
  Change in self-transcendent state will be measured with the Nondual Awareness Dimensional Assessment - State Version. Scores range from 0 to 10, with higher scores reflecting greater self-transcendence.
Perceived Discrimination | Baseline, post treatment (one week after the final treatment session), and follow-up (one month after the final treatment session).
  Changes in the perception of experiencing discrimination (Everyday Discrimination). Scores range from 0 -54 with higher scores indicating higher levels of discrimination.
Connectedness to Nature Questionnaire | Baseline, post treatment (one week after the final treatment session), and follow-up (one month after the final treatment session).
  The effects on Connectedness to Nature as a moderator between treatment and outcomes. The scale consists of 16 items rated on a 5-point Likert scale, from 1 (strongly disagree) to 5 (strongly agree) and is scored by creating a mean of the 16 items, with scores ranging from one to five, with higher scores indicating a stronger connectedness to nature than lower scores.
Dispositional Mindfulness Scale | Baseline, post treatment (one week after the final treatment session), and follow-up (one month after the final treatment session).
  The Metacognitive Processes of Decentering scale (MPoD-t) will be used to assess the effects of dispositional mindfulness as a moderator between treatment and outcomes. Scores range from 0-80 with higher scores indicating higher dispositional mindfulness.
Sense of Belonging in College | Baseline, post treatment (one week after the final treatment session), and follow-up (one month after the final treatment session).
  The role of treatment type on the participant's sense of belonging in college. Scores range from 0-56 with higher scores indicating higher levels of belonging.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Lecy, PhD, Principal Investigator — Assistant Professor
Locations (1):
- University of South Dakota, Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Steer RA, Brown GK, Beck AT, Sanderson WC. Mean Beck Depression Inventory-II scores by severity of major depressive episode. Psychol Rep. 2001 Jun;88(3 Pt 2):1075-6. doi: 10.2466/pr0.2001.88.3c.1075. PMID 11597055
- [Background] Hanley AW, Garland EL. Mapping the Affective Dimension of Embodiment With the Sensation Manikin: Validation Among Chronic Pain Patients and Modification by Mindfulness-Oriented Recovery Enhancement. Psychosom Med. 2019 Sep;81(7):612-621. doi: 10.1097/PSY.0000000000000725. PMID 31246748
- [Background] Hanley AW, Nakamura Y, Garland EL. The Nondual Awareness Dimensional Assessment (NADA): New tools to assess nondual traits and states of consciousness occurring within and beyond the context of meditation. Psychol Assess. 2018 Dec;30(12):1625-1639. doi: 10.1037/pas0000615. Epub 2018 Jul 30. PMID 30058824
- [Background] Knowles KA, Olatunji BO. Specificity of trait anxiety in anxiety and depression: Meta-analysis of the State-Trait Anxiety Inventory. Clin Psychol Rev. 2020 Dec;82:101928. doi: 10.1016/j.cpr.2020.101928. Epub 2020 Oct 10. PMID 33091745
- [Background] Sims M, Wyatt SB, Gutierrez ML, Taylor HA, Williams DR. Development and psychometric testing of a multidimensional instrument of perceived discrimination among African Americans in the Jackson Heart Study. Ethn Dis. 2009 Winter;19(1):56-64. PMID 19341164
- [Background] Felitti VJ, Anda RF, Nordenberg D, Williamson DF, Spitz AM, Edwards V, Koss MP, Marks JS. Relationship of childhood abuse and household dysfunction to many of the leading causes of death in adults. The Adverse Childhood Experiences (ACE) Study. Am J Prev Med. 1998 May;14(4):245-58. doi: 10.1016/s0749-3797(98)00017-8. PMID 9635069
- [Background] Navarro O, Olivos P, Fleury-Bahi G. "Connectedness to Nature Scale": Validity and Reliability in the French Context. Front Psychol. 2017 Dec 12;8:2180. doi: 10.3389/fpsyg.2017.02180. eCollection 2017. PMID 29312052